CLINICAL TRIAL: NCT03514160
Title: Does Exercise-induced Improvements in Emotion Regulation Enhance Daily Physical Activity and Well-being in Frail Sedentary Older Adults?
Brief Title: Relationships Between Exercise and Emotion Regulation on Physical Activity in Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: G00004606
Record Dates: First submitted 2017-04-07; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-04

CONDITIONS: Mobility Limitation; Sedentary Lifestyle; Older Adults
MeSH Terms: conditions — Mobility Limitation; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomization to group exercise or an attention-control group for 12 weeks (2:1 ratio). Group exercise sessions took place once per week at a community center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group exercise (Active Comparator): Group exercise training at a community site. Exercises included supervised upper and lower-body strength and balance exercises twice per week. Hand-made, weighted bars were used for resistance props and balance. The exercises included: chair squats; standing single leg hip abduction; hip extension; balance heal-to-toe walking; seated hip adduction and knee extension; wall push-ups; bent-over rows; shoulder press; elbow flexion and extension).
  Interventions: Behavioral: Group exercise
- Attention-Control group (No Intervention): Attendance to community site usual activities offered to older adults. Participants in this group were offered the exercise routine after completing the 12-week study.

INTERVENTIONS:
Behavioral: Group exercise — Group exercise based on the American College of Sports Medicine guidelines.
  Arms: Group exercise

SUMMARY:
Frailty in older adults is a consequence of physical inactivity, which leads to poor physical function, disability and poor health outcomes. Nearly 60% of older adults report inactivity. Emotion regulation strategies have affective, cognitive and social consequences. Positive emotions are significantly associated with a higher ability to perform activities of daily living. There is a gap in the understanding of how exercise influences the selection of emotion regulation strategies (avoidant vs. adaptive) in frail older adults. The investigators propose to examine the interactions between regular exercise, selection of emotional regulation strategies, and daily physical activity in frail sedentary older adults.

DETAILED DESCRIPTION:
1. Determine the choice of emotion regulation strategies used by frail sedentary older adults (60+ years; n=24). Frailty will be defined as a gait speed <0.8 m/sec.

   Hypothesis: Frail sedentary older adults will choose avoidant emotion regulation strategies.
2. Examine whether a peer-led, community-based, group-exercise program lasting 12-weeks improves the selection of emotion regulation strategies in frail sedentary older adults as compared to those receiving support services (12/group).

   Hypothesis: Exercise will result in higher use of adaptive emotion regulation strategies than support services.
3. Examine if improved selection of emotional regulation strategies with exercise translates into increased daily physical activity and reduced sedentary behavior by frail older adults as compared to those receiving support services.

   Hypothesis: Exercise will significantly increase daily physical activity and decrease sedentary behavior than support services.
4. Determine if improvements in emotional regulation strategy selection and daily physical activity levels positively influence health and well-being (i.e. health status, physical function, mood, depressive symptoms, anxiety, and sense of loneliness and isolation).

Hypothesis: Exercise-induced improvements in emotion regulation and increased daily physical activity will be associated with improved overall health and well-being as compared to support services.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults 60+ years of age
* Men and women
* Frail older adults with impaired mobility (gait speed < 0.8 m/sec)
* Sedentary older adults

Exclusion Criteria:

* Unable to give consent
* Unable to exercise
* Unable to travel to the community site
* Unstable chronic conditions

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Seven-day free living physical activity | 12 weeks
  Number of steps per day were objectively measured with an activity monitor worn for a seven-day period

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Castaneda-Sceppa, MD, PhD, Principal Investigator — Professor and Chair
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No